CLINICAL TRIAL: NCT05879718
Title: A PHASE 2, DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED, MULTICENTER STUDY TO EVALUATE THE CLINICAL EFFECT, PHARMACODYNAMIC, PHARMACOKINETIC AND SAFETY PROFILE OF PF 06823859 IN ADULT PARTICIPANTS WITH ACTIVE CLE OR SLE WITH CUTANEOUS MANIFESTATIONS
Brief Title: A Study to Learn About the Study Medicine (PF-06823859) in Adults With Active CLE or SLE With Skin Symptoms.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Pfizer has made an internal business decision to not continue this study. This decision was not due to safety concerns or clinical effect reasons or requests from any regulatory authorities.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C0251013; 2023-503343-33-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Lupus Erythematosus, Systemic; Lupus Erythematosus, Cutaneous
Keywords: type 1 IFN gene signature, SLE, CLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Intervention Model Description: About 48 eligible participants will be randomized in a 2:1 ratio to receive either PF-06823859 or placebo. Following assessments for the primary endpoint at Week 12, participants who are receiving active PF-06823859 or who are placebo non responders (responder is defined by ≥4 point reduction from the baseline in CLASI-A score) will receive PF-06823859 beginning at Week 16, while placebo responders will continue to be in the placebo group. The last dose of study intervention will be administered at Week 40 followed by last full study assessments at Week 48. The final follow up visit will be conducted at Week 60.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): PF-06823859
  Interventions: Drug: PF-06823859
- Group 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo (intravenous infusion)
  Arms: Group 2
Drug: PF-06823859 — PF-06823859 (intravenous infusion)
  Arms: Group 1

SUMMARY:
The purpose of this study is to learn about the effects, safety and how PF-06823859 is processed in adults with cutaneous lupus erythematosus (CLE) or systemic lupus erythematosus (SLE) showing some skin symptoms.

This study is seeking for participants who:

* are adults of 18 years of age or older.
* are confirmed to have CLE or SLE with involvement of the skin.
* have a Cutaneous Lupus Erythematosus Disease Area and Severity Index activity (CLASI-A) score of at least 8.

About 48 participants will be selected to receive active study medicine (PF-06823859) or placebo (an infusion without drug). About 32 are grouped to receive the active study medicine and 16 are to receive placebo. They will be receiving the treatments by intravenous infusion (injected directly into the veins).

At week 16 all participants receiving the active study drug since day 1 and participants who have received placebo since day 1 and are not responding clinically will receive active study medication. Patients who have received placebo since Day 1 and who have had a clinical response will continue to receive placebo till week 40. All participants will have last follow-up visit at Week 60.

The study will compare participants receiving PF-06823859 to participants who receive placebo. This will help us see if PF-06823859 is safe and effective to treat CLE or SLE with skin symptoms and improve participant's CLASI-A score. Participants will take part in this study for about 65 weeks. This includes up to a 5-week selection period, a 12-week Q4Wk treatment period, a 36-week Q8Wk treatment period, and a 12-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically confirmed active CLE or SLE with cutaneous manifestations in the form of subacute cutaneous lupus erythematosus or/and discoid/chronic cutaneous lupus erythematosus at least 3 months and CLASI-A at least 8 or higher.
* Participant has adequate intravenous infusion access per investigator's judgement
* Willing to comply with study procedures including skin punch biopsies procedures.
* Weight is greater than 40 kg and less than 130 kg.

Exclusion Criteria:

* Skin disorders other than CLE or SLE.
* Active, severe lupus nephritis requiring treatment with cytotoxic agents or high-dose steroids.
* Active severe central nervous system lupus requiring therapeutic intervention within 60 days of baseline.
* Cancer or a history of cancer within 5 years of screening except adequately resected basal or squamous cell carcinoma of the skin, or carcinoma in situ of uterine cervix.
* Known history of a major cardiovascular or cerebrovascular event within 24 months, pulmonary arterial hypertension, pulmonary embolism within 6 months of screening.
* Have any autoimmune or inflammatory disease that would interfere with interpretation of test results or clinical assessments.
* History of disseminated herpes zoster/simplex or recurrent herpes zoster.
* Serious infection within 60 days of baseline or an active infection treated with oral antibiotics within 14 days of baseline.
* Have evidence of active or latent infection of hepatitis B or C, known history of human immunodeficient virus (HIV) infection, or infected with Mycobacterium TB (active or latent TB)
* Laboratory abnormalities that meet exclusion criteria at the Screening visit. The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in type 1 IFN GS score in lesional skin at Week 12 | Week 12
  A 13-gene IFN gene signature score was used to measure IFN activity at both baseline and week 12, the gene signature score is assessed per sample by averaging the log2CPM(Counts Per Million reads) values of these 13 genes through RNAseq profiling. The gene signature score is positively linked to the gene expression activity of those 13 genes that are related to IFN.

SECONDARY OUTCOMES:
Percent change from baseline in CLASI-A score at Week 12 | Week 12
  The Cutaneous Lupus Erythematosus Disease Activity and Damage Score
Percent change from baseline in CLASI-A (over time in addition to Week 12) | Week 4, 8, 12, 16, 20, 24, 32, 40, 48, and 60
  Percent Change from Baseline in Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity (CLASI-A) Score
Change from baseline in CLASI-A score (over time) | Week 4, 8, 12, 16, 20, 24, 32, 40, 48, and 60
  Change from Baseline in Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity (CLASI-A) Score
Achieving ≥50%, 4 or 7 points reduction in CLASI-A (over time) | Week 4, 8, 12, 16, 20, 24, 32, 40, 48, and 60
  Achieving ≥50%, 4 or 7 points reduction in CLASI-A
Change from baseline in Physician global assessment (PhGA) (over time) | Week 4, 8, 12, 16, 20, 24, 32, 40, 48, and 60
  The PhGA is a visual analog scale (VAS) tool to measure worsening in the participant general health status. Physician will place a mark on the scale between 0 (none), 1 (mild), 2(moderate) and 3 (severe).
Incidence and severity of laboratory, vital signs, 12-lead ECG abnormalities, AEs, SAEs and withdrawals due to AEs over time | Day 1, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 56, and 60

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- United States (11):
  - The Kirklin Clinic of UAB Hospital, Birmingham, Alabama
  - University of Alabama at Birmingham - School of Medicine, Birmingham, Alabama
  - University of Alabama at Birmingham, Department of Dermatology, Birmingham, Alabama
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic in Arizona - Scottsdale, Scottsdale, Arizona
  - Dermatology Research Associates, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - The University of Kansas Hospital, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cleveland Clinic Foundation, Cleveland, Ohio
- Canada (3):
  - DermEffects, London, Ontario
  - Dermatology on Bloor - Research Toronto, Toronto, Ontario
  - Whitby Health Centre, Whitby, Ontario
- Greece (3):
  - University General Hospital "ATTIKON" - General Hospital of West Attica "H AGIA VARVARA", Chaïdári, Attikí
  - Ionos Dragoumi 5 Kaisariani, Kaisarianí, Attikí
  - Dermatological and Venereological Hospital Andreas Syggros, Athens
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0251013